CLINICAL TRIAL: NCT03355677
Title: A Clinical Interventional Study Into Airways Disease Case Finding and Complex Case Management
Brief Title: A Study Into Airways Disease Case Finding and Management
Acronym: ASSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University Hospital Southampton NHS Foundation Trust (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CLAHRC 001
Record Dates: First submitted 2017-01-13; First posted 2017-11-28 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: COPD; Asthma
Keywords: Case finding; complex case management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Intervention Model Description: All patient identified by an electronic algorithm as at risk of having possible COPD were invited to attend a case finding clinic at their local GP practice for lung function testing. The algorithm was applied to control group practices and the number of new cases of COPD in the records was compared. 'At risk' patients with existing asthma and COPD were also invited to attend, and have their health status reviewed. We were unable to complete control group comparisons on this group of patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Case finding clinics (Active Comparator): The visit will be a minimum 90 minutes long at the participants own GP surgery. This will include a respiratory assessment including spirometry will performed by a RT Respiratory Nurse Specialist (RNS) and where possible a Practice Nurse or Nurse Practitioner will attend. The visit will consist of objective measurements, investigations and questionnaires
  Interventions: Procedure: Case finding Clinic
- Case finding Usual care (Placebo Comparator): In the control arm of the study, practices will continue with usual care according to national guidance for case finding for COPD (NICE, 2010). Matched practices will have their eligible population identified through electronic searches based on data routinely recorded in primary care run in the HHRa. Case finding yield will be measured as the percentage of patients from the eligible population identified with a respiratory diagnosis in the 12 months from study beginning to study end.
  Interventions: Other: Usual Care
- At Risk Case clinics (Active Comparator): The complex case clinic will be a minimum 120 minute appointment at the participants own GP surgery. The intervention will include an initial assessment by a RT Respiratory Nurse Specialist (RNS) and followed by a joint assessment by a respiratory physician (RP) working alongside a practice clinician (GP and/or Practice Nurse/Nurse Practitioner). The visit will consist of objective measurements, investigations and questionnaires as outlined in section 3 below. A personalised disease management and action plan will be agreed jointly between the RT, practice clinician and participant. The practice clinician will undertake the necessary tasks required for the agreed management plan. The clinical responsibility for the participant will remain with the GP practice.
  Interventions: Procedure: At Risk Case Clinics
- At Risk Usual Care (Placebo Comparator): In the control arm of the study, practices will continue with usual care according to national guidance for the management of COPD and asthma . A cohort of patients matched for practice and for age, sex, disease condition and, where possible, disease control will be identified. This cohort will be monitored against markers of sub-optimal disease (medication usage, exacerbations, unscheduled visits to the practice, attendance or admission to hospital).
  Interventions: Other: Usual Care

INTERVENTIONS:
Procedure: Case finding Clinic — Case finding clinic - participants will be reviewed by a respiratory specialist team. Full respiratory history will be taken and physical examination will be preformed. The participant will then complete 3 quality of life and functionality questionnaires the MRC dyspnoea score and the COPD diagnostic questionnaire. They will then be asked to perform FeNO CO and spirometry measurements.
  Arms: Case finding clinics
Procedure: At Risk Case Clinics — Complex Case Clinic participants will be reviewed by a respiratory specialist team. Full respiratory history will be taken and physical examination will be preformed. The participant will then complete 6 quality of life and functionality questionnaires . They will then be asked to perform FeNO CO and spirometry measurements. Participants inhaler technique will be checked and any errors corrected. Smoking cessation advice and support will be given if necessary. Each participant will be given an individualised self management plan.
  Arms: At Risk Case clinics
Other: Usual Care — The control surgeries selected by the HHRA will continue with usual care.
  Arms: At Risk Usual Care; Case finding Usual care

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a disease of the lungs which is generally caused by smoking tobacco. It is a largely preventable disease that causes severe and irreversible damage to the lungs. If not detected early, this damage will progress causing significant breathing difficulties, disability and poor survival rates. Patients with COPD can experience exacerbations of their disease which can also lead to can be described as a worsening of the patients symptoms COPD is a global health concern and it is estimated to become the third leading cause of death by 2020. In the United Kingdom, around 900,000 people have a formal diagnosis of COPD. However, it is believed that over 2 million more people may be living with the disease and are unaware that they have it. The cost of treating lung disease in the National Health Service (NHS) is estimated to be approximately £4.7billion per year . The majority of these costs are caused by a small group of COPD patients with severe disease and complex problems , . Late diagnosis has been proven as a contributing factor to the worsening of COPD, disease progression and increased healthcare costs. Indeed, recent research has shown that patients may attend their general practitioner (GP) practice with signs of the disease up to five years before they have the condition diagnosed. A delay in diagnosis is known to hasten the decline in lung function and worsen disease severity making treatment options less useful in the long term. This has led to national guidelines recognising that patients with COPD need to be diagnosed and treated effectively at the earliest opportunity.

The aim of this study is to find the best way to identify or 'case find' patients who have not yet been diagnosed with COPD, and also identify patients with more complex disease using a computerised search programme. The study will examine whether this intervention has saved the NHS money by reducing GP and hospital visits and by decreasing rescue medicine usage for respiratory problems, by comparing this data to similar GP practices where the intervention had not been implemented. Once patients have been identified, they will be invited to attend a clinic appointment at their GP practice to participate in a tailored intervention programme for patients at risk of having COPD and those with existing complex COPD. GP practices will also be offered a training package in order to continue the intervention programme in the future.

DETAILED DESCRIPTION:
Background Chronic Obstructive Pulmonary Disease (COPD) COPD is a disease of the lungs characterised by airway inflammation leading to airflow obstruction. It is a progressive and largely preventable disease caused by the inhalation of noxious gases generally through cigarette smoking. Patients experience persistent symptoms including breathlessness, reduced exercise tolerance and an increase in the production of mucus in the airways. The impact of the disease to the individual is substantial in terms of physical disability and psycho-social issues.

Patients with COPD can experience an exacerbation of their disease, defined as a sudden worsening of symptoms above and beyond the individual's normal daily variation. COPD exacerbations are the second most common cause of emergency hospital admissions in the UK, with an estimated 94,000 admissions per annum. Indeed, COPD is one of the most expensive inpatient conditions in the UK, costing the National Health Service (NHS) over £800 million in direct healthcare costs. COPD is also set to become the third leading cause of death worldwide by the year 2030, surpassed only by heart disease and stroke. Despite this high level of mortality, public awareness of COPD is low in the United Kingdom (UK): around 89% of the general public have never heard of COPD.

Under-diagnosis of COPD Evidence suggests that 13% of people over 35 have COPD but many are diagnosed late and most are currently undiagnosed. Almost a third of patients admitted to hospital with a COPD exacerbation had not been diagnosed. Opportunities for early diagnosis of COPD are missed in primary care: a recent study demonstrated that 85% of patients had consulted primary care with lower respiratory symptoms in the five years immediately before their diagnosis of COPD. The insidious onset of COPD means undiagnosed patients may unconsciously modify their way of life, and only present to primary care in the later stages of disease. Furthermore, smokers, who constitute a substantial portion of the target population for case finding, have been shown to hold self-exempting beliefs and thus may be less likely to present to primary care. In addition, many patients visit their GP for problems related to COPD, such as chest infections and breathlessness, but the correct diagnosis is not made.

The importance of early diagnosis of COPD National health policy initiatives in the UK underscore improved diagnosis as a priority Early diagnosis of COPD followed by optimisation of treatment has potential cost savings for the NHS of more than £1 billion over 10 years . Prevention strategies (smoking cessation, dietary, exercise promotion, self-management and vaccination) can be targeted on this group of patients to maintain and improve health, and appropriate pharmacologic therapies (that can improve symptoms, exercise tolerance and quality of life and reduce the risk of exacerbations) commenced in newly identified people if appropriate. A recent systematic review of the literature concluded that a combination of a screening questionnaire and micro-spirometry seems to demonstrate the best overall screening test accuracy, but there has been little uptake of this strategy in UK primary care and doubts remain as to its feasibility and cost-effectiveness. However, whilst a variety of approaches to case finding have been trialled world-wide published studies have been variable in quality and the most effective, economical method of screening has yet to be identified. The National Institute for Health and Clinical Excellence (NICE) and the Department of Health (DoH) in the UK have recommended both systematic and opportunistic case finding to diagnose symptomatic patients . The UK National Screening Committee concurs, explicitly recommending case finding (defined as targeting patients with symptoms suggestive of COPD) rather than screening (defined as identifying apparently healthy people who may be at increased risk of COPD). A recent All Party Parliamentary Group report on Respiratory Deaths (APPG RD) concluded that tools to aid health care professionals to case find for COPD need to be developed in order to prioritise for use at national level.

Case-finding: identifying symptomatic but not yet diagnosed patients 'TargetCOPD' is an ongoing NIHR funded randomised controlled trial comparing the cost-effectiveness of two alternative case-finding approaches for identifying undiagnosed COPD. Both approaches rely on patient self-reported questionnaires to identify symptoms; one opportunistically administered, the other systematically administered. 'TargetCOPD' should provide some useful information on case-finding using questionnaires. However, evidence suggests that alternative approaches to case finding such as electronic searches based on routine primary care data may be a valuable tool for identifying symptomatic patients with as yet undiagnosed COPD. However, further validation of electronic case-finding strategies is required.

In early 2015 the Wessex CLAHRC, WAHSN and West Hampshire CCG ran a service development project in two surgeries in West Hampshire using notes review and a different electronic case finding instrument, GRASP-COPD. The project identified a need for further investigation into the efficiency of case-finding strategies.

The investigators propose to use an electronic case-finding algorithm developed and validated in Birmingham, UK as part of a NIHR funded programme grant centred on case finding for COPD.

'Complex' patients: identification and management Over the past two decades, there has been a shift in the locus of care for the majority of patients with chronic respiratory diseases in the UK towards the community. Respiratory diseases are amongst the most common causes of primary care consultations, accounting for 24 million consultations annually. Increasing numbers of complex respiratory patients are being managed in the primary care setting by generalist teams, with a focus on avoidance of admissions to hospital. Specialist secondary care is restricted to those patients admitted to hospital in a crisis or referred because of uncontrolled disease.

There is evidence of significant and unwarranted variability in the standards of respiratory management in both the primary and secondary care sectors. Marked variations in outcomes for patients with respiratory disease have also been shown, both regionally and between individual General Practitioner (GP) practices. There is evidence linking the quality of care provided in general practice with unplanned admissions to secondary care , and decreased admission rates have been reported in a number of long-term conditions (including COPD and asthma) where GPs were financially incentivised to provide high-quality care . Moreover, higher levels of professional education, nurse staffing and clinical recording in primary care are all associated with an improvement in the quality of clinical care for patients with COPD. However, a 'skills gap' may exist in some primary care settings, where GPs and other health care professionals lack advanced training in the management of these common conditions, particularly in the case of patients with multi-morbidity, uncertain diagnosis or complex problems .

The investigators have performed pilot studies which have identified widespread variability in practice level competencies for the diagnosis and management of respiratory conditions in primary care; in particular quality assured spirometry is only performed in a minority. No practices currently deliver FeNO measurements central to draft NICE Asthma guidelines. Knowledge of inhaled therapy options and techniques is highly variable. Patients with more severe or complicated disease may receive suboptimal care, which may in turn lead to poor outcomes. Such patients may fail to reach a specialist assessment that could potentially improve outcomes, either because they are not offered referral to a specialist clinic or because they decline going to a hospital clinic for such an assessment. Therefore, a community-based integrated care approach with joint specialist-generalist "mentorship" clinics in the community which utilise both specialist skills and the overall holistic perspective of the generalist primary care teams may be a promising solution. We have piloted a series of such 'mentorship' clinics as part of a service improvement programme of work with West Hampshire Clinical Commissioning Group (WHCCG) and the Wessex Academic Health Sciences Network (WAHSN). Pilot data suggest significant impacts on suboptimal outcomes including a reduction in inappropriate inhaled medication, exacerbations, unscheduled visits to primary care and attendance and admission to hospital. Furthermore, attendance rates and feedback from patients and care-givers suggest such clinics have high levels of acceptability to patients and their families.

Further potential benefits of 'mentorship' clinics in the community include not only improvement in quality of care for each of the individual patients seen, but also on-site education for the primary care teams, leaving a legacy of improved skills and greater confidence in managing complex disease. Such clinics have the potential to increase patient and staff satisfaction, reduce secondary care use and consequently reduce the financial burden of respiratory disease on the local health economy.

Up to 20 GP practices throughout Wessex will be recruited to the intervention arm. Practices in the intervention arm will be recruited pragmatically through the relevant CCG or local clinical and academic networks. Practices will be supported by the clinical research team from study set up to study end. The study team will directly engage with each practice in order to ensure that study processes align with administrative and clinical arrangements in each specific practice. A briefing/debriefing session will be held with each practice prior to the study commencing and at study conclusion.

Practices in the control arm will be matched if possible by size, demographic profile, socio-economic status profile and rural/urban setting. Control practices will be identified through the Hampshire Health Record Analytic Database (HHRA). The HHRA is a separate electronic database created for research, analysis and commissioning support within the local NHS. It currently includes data from 133 practices across Hampshire which is linked to the GP patient database system. The Governance body is the Hampshire Health Record Advisory Group (HHRAG), which ensures the security and confidentiality of the HHRA and HHR (Hampshire Health Records) and considers issues of data integration, data sharing and data extraction/analysis. The HHRA receives data monthly from the HHR, but in a pseudonymised format,. Although the HHRA can be viewed in a pseudonymised format by analysts working directly with the database, all data used for research purposes is extracted in an anonymised format.

ELIGIBILITY:
Inclusion Criteria: Case Finding

* • Registered with one of the participating GP practices as at 1st January 2015

  * ≥40 years old
  * Ex or current smoker
  * No COPD diagnosis
  * Willing and able to give written informed consent.

Exclusion Criteria:

* • Unable to give informed consent

  * Suffering from a terminal illness
  * Patients whom the GP or clinical investigator deem inappropriate to participate
  * Existing COPD diagnosis
  * Obvious contraindications to spirometry (e.g. unstable abdominal aortic aneurysm)
  * Under secondary care for investigation of breathlessness
  * Pregnant
  * Housebound

Inclusion Criteria - Complex Case Management

* Registered with one of the participating GP practices as at 1st January 2015
* On the practice COPD or asthma registers
* Identified by the electronic search Exclusion Criteria
* Unable to give informed consent
* Suffering from a terminal illness
* Patients whom the GP or clinical investigator deem inappropriate to participate
* No existing respiratory diagnosis
* Under secondary care for respiratory issues
* Housebound

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2017-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Case finding | 12 months
  The proportion of those patients identified by the case-finding algorithm at the chosen threshold who are diagnosed with COPD within 12 months following assessment at a case-finding clinic (for the intervention group practices) or following the practice-matched index date (for the control group practices). For the intervention group this will be the proportion of those invited to attend. For the control group this will be the proportion of those patients who would have been invited to attend, based on identical case-finding algorithm criteria.

SECONDARY OUTCOMES:
Attendance - Case finding | 12 months
  The proportion of all patients identified by Read code algorithm in intervention practices compared to matched practices in the control group who attend case finding clinics
Newly Diagnosed - Case finding | 12 months
  The proportion of all patients identified by Read code algorithm in intervention practices compared to matched practices in the control group who • Are newly diagnosed with asthma, COPD or other respiratory disorder or have a change in diagnosis made.
Co Morbidities - case finding | 12 months
  The proportion of all patients identified by Read code algorithm in intervention practices compared to matched practices in the control group who• Have additional co-morbidities identified.
Treatments - case finding | 12 months
  The proportion of all patients identified by Read code algorithm in intervention practices compared to matched practices in the control group who • Have new treatment commenced, including changes to prescribed medication and non-pharmacological interventions initiated
Smoking cessation - case finding | 12 months
  The proportion of all patients identified by Read code algorithm in intervention practices compared to matched practices in the control group who • Are referred on to smoking cessation services, and succeed in quitting smoking.
secondary care referrals - case finding | 12 months
  The proportion of all patients identified by Read code algorithm in intervention practices compared to matched practices in the control group who require referral on to secondary care
smoking - | 12 months
  proportion of patients who are referred on to smoking cessation services, and succeed in quitting smoking
Broncholdilator Usage | 12 months
  Number of prescribed short acting bronchodilators administered to patients
Corticosteroids | 12 months
  number of prescribed episodes of oral coticosteroids
Healthcare Usage | 12 months
  Number of episodes of Health care usage utilised by patient
Breathlessness | 6 and 12 mths
  improvement in Breathlessness scores recorded by patients using the Medical Research Council breathlessness score. Grading from 1-5 to establish clinical grade of breathlessness on daily activity. Higher values are considered to mean greater impact on functionality.
Anxiety | 6,12 months
  anxiety scores recorded by patients using the GAD7 questionnaires
Healthcare status | 6,12 months
  improvements in Healthcare status using EQ 5D questionnaire
Airway disease control | 6,12 months
  improvement in disease control using the COPD Assessment Test
Admission | 12 months
  Proportion of Emergency Department and hospital admissions
Exacerbations | 12 months
  proportion of exacerbations experienced by patients
Depression | 6,12 months
  Depression scores recorded by patients using the PHQ9 questionnaires
Asthma disease control | 6,12 months
  improvement in disease control using Asthma Control Test
COPD Severity | 6,12 months
  improvements in Healthcare status using DOSE
Primary care attendance | 12 months
  Comparison of the primary care attendance rate among the group of patients attending the 'at risk' in the year before clinic attendance with the year after.
Number of respiratory consultations | 12 months
  Comparison of the respiratory consultation rate in primary care among the cohort of patients invited for a complex case review (i.e. attendance at the 'at risk' clinic) with a comparator cohort of patients identified as being 'at risk' within a group of practices matched to the 'at risk' intervention group of practices.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wilkinson, Study Director — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anthonisen NR, Manfreda J, Warren CP, Hershfield ES, Harding GK, Nelson NA. Antibiotic therapy in exacerbations of chronic obstructive pulmonary disease. Ann Intern Med. 1987 Feb;106(2):196-204. doi: 10.7326/0003-4819-106-2-196. PMID 3492164
- [Background] Badia X, Schiaffino A, Alonso J, Herdman M. Using the EuroQoI 5-D in the Catalan general population: feasibility and construct validity. Qual Life Res. 1998 May;7(4):311-22. doi: 10.1023/a:1024933913698. PMID 9610215
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Busby J, Purdy S, Hollingworth W. A systematic review of the magnitude and cause of geographic variation in unplanned hospital admission rates and length of stay for ambulatory care sensitive conditions. BMC Health Serv Res. 2015 Aug 13;15:324. doi: 10.1186/s12913-015-0964-3. PMID 26268576
- [Background] Dang-Tan T, Ismaila A, Zhang S, Zarotsky V, Bernauer M. Clinical, humanistic, and economic burden of chronic obstructive pulmonary disease (COPD) in Canada: a systematic review. BMC Res Notes. 2015 Sep 21;8:464. doi: 10.1186/s13104-015-1427-y. PMID 26391471
- [Background] Dirven JA, Tange HJ, Muris JW, van Haaren KM, Vink G, van Schayck OC. Early detection of COPD in general practice: patient or practice managed? A randomised controlled trial of two strategies in different socioeconomic environments. Prim Care Respir J. 2013 Sep;22(3):331-7. doi: 10.4104/pcrj.2013.00070. PMID 23966214
- [Background] Jordan RE, Adab P, Sitch A, Enocson A, Blissett D, Jowett S, Marsh J, Riley RD, Miller MR, Cooper BG, Turner AM, Jolly K, Ayres JG, Haroon S, Stockley R, Greenfield S, Siebert S, Daley AJ, Cheng KK, Fitzmaurice D. Targeted case finding for chronic obstructive pulmonary disease versus routine practice in primary care (TargetCOPD): a cluster-randomised controlled trial. Lancet Respir Med. 2016 Sep;4(9):720-730. doi: 10.1016/S2213-2600(16)30149-7. Epub 2016 Jul 19. PMID 27444687
- [Background] Foundation BL. Lung disease in the UK - big picture statistics 2016 [Available from: https://statistics.blf.org.uk/lung-disease-uk-big-picture.
- [Background] Foundation BL. Asthma Statistics 2016 [Available from: https://statistics.blf.org.uk/asthma.
- [Background] Foundation BL. Chronic obstructive pulmonary disease (COPD) Statistics 2016 [Available from: https://statistics.blf.org.uk/copd.
- [Background] Gibson GJ, Loddenkemper R, Lundback B, Sibille Y. Respiratory health and disease in Europe: the new European Lung White Book. Eur Respir J. 2013 Sep;42(3):559-63. doi: 10.1183/09031936.00105513. No abstract available. PMID 24000245
- [Background] Bateman ED, Hurd SS, Barnes PJ, Bousquet J, Drazen JM, FitzGerald JM, Gibson P, Ohta K, O'Byrne P, Pedersen SE, Pizzichini E, Sullivan SD, Wenzel SE, Zar HJ. Global strategy for asthma management and prevention: GINA executive summary. Eur Respir J. 2008 Jan;31(1):143-78. doi: 10.1183/09031936.00138707. PMID 18166595
- [Background] Levy ML. National Review of Asthma Deaths (NRAD). Br J Gen Pract. 2014 Nov;64(628):564. doi: 10.3399/bjgp14X682237. No abstract available. PMID 25348975
- [Background] Department of Health. A Outcomes Strategy for people with Chronic Obstructive Pulmonary Disease and Asthma in England. 2011.
- [Background] Asthma UK. Living on a Knife Edge. 2003
- [Background] ten Brinke A, Sterk PJ, Masclee AA, Spinhoven P, Schmidt JT, Zwinderman AH, Rabe KF, Bel EH. Risk factors of frequent exacerbations in difficult-to-treat asthma. Eur Respir J. 2005 Nov;26(5):812-8. doi: 10.1183/09031936.05.00037905. PMID 16264041
- [Background] Chung KF BE, Wenzel ES, . Difficult-to-treat severe asthma. 2011 ed. Sheffield: ERS. p. 120-9.
- [Background] Moore WC, Bleecker ER, Curran-Everett D, Erzurum SC, Ameredes BT, Bacharier L, Calhoun WJ, Castro M, Chung KF, Clark MP, Dweik RA, Fitzpatrick AM, Gaston B, Hew M, Hussain I, Jarjour NN, Israel E, Levy BD, Murphy JR, Peters SP, Teague WG, Meyers DA, Busse WW, Wenzel SE; National Heart, Lung, Blood Institute's Severe Asthma Research Program. Characterization of the severe asthma phenotype by the National Heart, Lung, and Blood Institute's Severe Asthma Research Program. J Allergy Clin Immunol. 2007 Feb;119(2):405-13. doi: 10.1016/j.jaci.2006.11.639. PMID 17291857
- [Background] Global Initiative for Chronic Obstructive Lung Disease. Global starergy for the diagnosis, management and prevention of chronic obstructive pulmonary disease, 2015 [Available from: http://www.goldcopd.it/materiale/2015/GOLD_Pocket_2015.pdf.
- [Background] Chronic obstructive pulmonary disease in over 16s: diagnosis and management. London: National Institute for Health and Care Excellence (NICE); 2019 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK542426/ PMID 31211541
- [Background] O'Donnell DE, Parker CM. COPD exacerbations . 3: Pathophysiology. Thorax. 2006 Apr;61(4):354-61. doi: 10.1136/thx.2005.041830. PMID 16565268
- [Background] All Party Palimentary Group on Respiratory Health. Report on the Inquiry into Respiratory Deaths 2014. Available from: https://www.blf.org.uk/take-action/campaign-with-us/appg-on-respiratory-health.
- [Background] World Health Organisation. Chronic obstructive pulmonary disease (COPD) 2004 [Available from: http://www.who.int/respiratory/copd/en/.
- [Background] British Lung Foundation. Invisible Lives. Chronic obstructive pulmonary disease (COPD) finding the missing millions 2007 [Available from: www.blf.org.uk/publications/detail/Invisible-Lives-report.
- [Background] Jones RC, Price D, Ryan D, Sims EJ, von Ziegenweidt J, Mascarenhas L, Burden A, Halpin DM, Winter R, Hill S, Kearney M, Holton K, Moger A, Freeman D, Chisholm A, Bateman ED; Respiratory Effectiveness Group. Opportunities to diagnose chronic obstructive pulmonary disease in routine care in the UK: a retrospective study of a clinical cohort. Lancet Respir Med. 2014 Apr;2(4):267-76. doi: 10.1016/S2213-2600(14)70008-6. Epub 2014 Feb 13. PMID 24717623
- [Background] Pinnock H, Kendall M, Murray SA, Worth A, Levack P, Porter M, MacNee W, Sheikh A. Living and dying with severe chronic obstructive pulmonary disease: multi-perspective longitudinal qualitative study. BMJ Support Palliat Care. 2011 Sep;1(2):174-83. doi: 10.1136/bmjspcare.d142rep. PMID 24653231
- [Background] Kotz D, Vos R, Huibers MJ. Ethical analysis of the justifiability of labelling with COPD for smoking cessation. J Med Ethics. 2009 Sep;35(9):534-40. doi: 10.1136/jme.2009.029280. PMID 19717691
- [Background] Department of Health. An outcomes strategy for people with chronic obstructive pulmonary disease (COPD) and asthma in England 2011 [Available from: https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/213840/dh_113279.pdf.
- [Background] Haroon SM, Jordan RE, O'Beirne-Elliman J, Adab P. Effectiveness of case finding strategies for COPD in primary care: a systematic review and meta-analysis. NPJ Prim Care Respir Med. 2015 Aug 27;25:15056. doi: 10.1038/npjpcrm.2015.56. PMID 26313400
- [Background] Riegels-Jakobsen T, Skouboe M, Dollerup J, Andersen CB, Staal LB, Jakobsen RB, Poulsen PB. Municipality screening of citizens with suspicion of chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2012;7:35-41. doi: 10.2147/COPD.S27314. Epub 2012 Feb 1. PMID 22315521
- [Background] Jordan RE, Lam KB, Cheng KK, Miller MR, Marsh JL, Ayres JG, Fitzmaurice D, Adab P. Case finding for chronic obstructive pulmonary disease: a model for optimising a targeted approach. Thorax. 2010 Jun;65(6):492-8. doi: 10.1136/thx.2009.129395. PMID 20522845
- [Background] Thorn J, Tilling B, Lisspers K, Jorgensen L, Stenling A, Stratelis G. Improved prediction of COPD in at-risk patients using lung function pre-screening in primary care: a real-life study and cost-effectiveness analysis. Prim Care Respir J. 2012 Jun;21(2):159-66. doi: 10.4104/pcrj.2011.00104. PMID 22270480
- [Background] Martinez FJ, Raczek AE, Seifer FD, Conoscenti CS, Curtice TG, D'Eletto T, Cote C, Hawkins C, Phillips AL; COPD-PS Clinician Working Group. Development and initial validation of a self-scored COPD Population Screener Questionnaire (COPD-PS). COPD. 2008 Apr;5(2):85-95. doi: 10.1080/15412550801940721. PMID 18415807
- [Background] Stanley AJ, Hasan I, Crockett AJ, van Schayck OC, Zwar NA. Validation of the COPD Diagnostic Questionnaire in an Australian general practice cohort: a cross-sectional study. Prim Care Respir J. 2014 Mar;23(1):92-7. doi: 10.4104/pcrj.2014.00015. PMID 24570082
- [Background] Frith P, Crockett A, Beilby J, Marshall D, Attewell R, Ratnanesan A, Gavagna G. Simplified COPD screening: validation of the PiKo-6(R) in primary care. Prim Care Respir J. 2011 Jun;20(2):190-8, 2 p following 198. doi: 10.4104/pcrj.2011.00040. PMID 21597667
- [Background] Sichletidis L, Spyratos D, Papaioannou M, Chloros D, Tsiotsios A, Tsagaraki V, Haidich AB. A combination of the IPAG questionnaire and PiKo-6(R) flow meter is a valuable screening tool for COPD in the primary care setting. Prim Care Respir J. 2011 Jun;20(2):184-9, 1 p following 189. doi: 10.4104/pcrj.2011.00038. PMID 21597666
- [Background] Kotz D, Nelemans P, van Schayck CP, Wesseling GJ. External validation of a COPD diagnostic questionnaire. Eur Respir J. 2008 Feb;31(2):298-303. doi: 10.1183/09031936.00074307. Epub 2007 Oct 24. PMID 17959636
- [Background] Haroon S, Adab P, Griffin C, Jordan R. Case finding for chronic obstructive pulmonary disease in primary care: a pilot randomised controlled trial. Br J Gen Pract. 2013 Jan;63(606):e55-62. doi: 10.3399/bjgp13X660788. PMID 23336474
- [Background] Jithoo A, Enright PL, Burney P, Buist AS, Bateman ED, Tan WC, Studnicka M, Mejza F, Gillespie S, Vollmer WM; BOLD Collaborative Research Group. Case-finding options for COPD: results from the Burden of Obstructive Lung Disease study. Eur Respir J. 2013 Mar;41(3):548-55. doi: 10.1183/09031936.00132011. Epub 2012 Jun 27. PMID 22743668
- [Background] Jordan RE, Adab P, Jowett S, Marsh JL, Riley RD, Enocson A, Miller MR, Cooper BG, Turner AM, Ayres JG, Cheng KK, Jolly K, Stockley RA, Greenfield S, Siebert S, Daley A, Fitzmaurice DA. TargetCOPD: a pragmatic randomised controlled trial of targeted case finding for COPD versus routine practice in primary care: protocol. BMC Pulm Med. 2014 Oct 4;14:157. doi: 10.1186/1471-2466-14-157. PMID 25280869
- [Background] Service TUNS. The UK NSC recommendation on Chronic Obstructive Pulmonary Disease 2013 [Available from: http://legacy.screening.nhs.uk/copd.
- [Background] Smith J HH, Edwards N, Maybin J, Parker H, Rosen R, Walsh N, . Securing the future of general practice: new models of primary care Nuffield Trust and King's Fund 2013 [updated 11/07/2016. Available from: http://www.nuffieldtrust.org.uk/sites/files/nuffield/publication/130718_securing_the_future_revised.pdf.
- [Background] Worth A, Pinnock H, Fletcher M, Hoskins G, Levy ML, Sheikh A. Systems for the management of respiratory disease in primary care--an international series: United Kingdom. Prim Care Respir J. 2011 Mar;20(1):23-32. doi: 10.4104/pcrj.2010.00070. PMID 21057735
- [Background] Harrison MJ, Dusheiko M, Sutton M, Gravelle H, Doran T, Roland M. Effect of a national primary care pay for performance scheme on emergency hospital admissions for ambulatory care sensitive conditions: controlled longitudinal study. BMJ. 2014 Nov 11;349:g6423. doi: 10.1136/bmj.g6423. PMID 25389120
- [Background] Levy ML. The national review of asthma deaths: what did we learn and what needs to change? Breathe (Sheff). 2015 Mar;11(1):14-24. doi: 10.1183/20734735.008914. PMID 26306100
- [Background] Griffiths P, Maben J, Murrells T. Organisational quality, nurse staffing and the quality of chronic disease management in primary care: observational study using routinely collected data. Int J Nurs Stud. 2011 Oct;48(10):1199-210. doi: 10.1016/j.ijnurstu.2011.03.011. Epub 2011 May 14. PMID 21571273
- [Background] Robertson et al. Specialist in out of hospital setting 2014 [updated http://www.kingsfund.org.uk/publications/specialists-out-hospital-settings.
- [Background] Asthma: diagnosis and monitoring of asthma in adults, children and young people. London: National Institute for Health and Care Excellence (NICE); 2017 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK469773/ PMID 29206391
- [Background] Evaluation of case finding for COPD/asthma and management of poorly controlled asthma/COPD project [Available from: http://wessexahsn.org.uk/img/projects/WHCCGWAHSNevaluation300415final%20(4).pdf
- [Background] Professor David Greenway. Shape of Training, Securing the future of excellent patient care 2013. Available from: http://www.shapeoftraining.co.uk/static/documents/content/Shape_of_training_FINAL_Report.pdf_53977887.pdf.
- [Background] Fletcher CM. Standardised questionniare on respiratory symptoms: a statement prepared and approved by the MRC commitee on the aetiology of chronic bronchitis (MRC breathlessness score) BMJ (Clinical research ed). 1960;2:1665.
- [Background] Mahler DA, Wells CK. Evaluation of clinical methods for rating dyspnea. Chest. 1988 Mar;93(3):580-6. doi: 10.1378/chest.93.3.580. PMID 3342669
- [Background] Pickard AS, Wilke C, Jung E, Patel S, Stavem K, Lee TA. Use of a preference-based measure of health (EQ-5D) in COPD and asthma. Respir Med. 2008 Apr;102(4):519-36. doi: 10.1016/j.rmed.2007.11.016. Epub 2008 Jan 3. PMID 18180151
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lamers F, Jonkers CC, Bosma H, Penninx BW, Knottnerus JA, van Eijk JT. Summed score of the Patient Health Questionnaire-9 was a reliable and valid method for depression screening in chronically ill elderly patients. J Clin Epidemiol. 2008 Jul;61(7):679-87. doi: 10.1016/j.jclinepi.2007.07.018. Epub 2008 Feb 14. PMID 18538262
- [Background] Phelan E, Williams B, Meeker K, Bonn K, Frederick J, Logerfo J, Snowden M. A study of the diagnostic accuracy of the PHQ-9 in primary care elderly. BMC Fam Pract. 2010 Sep 1;11:63. doi: 10.1186/1471-2296-11-63. PMID 20807445
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Swinson RP. The GAD-7 scale was accurate for diagnosing generalised anxiety disorder. Evid Based Med. 2006 Dec;11(6):184. doi: 10.1136/ebm.11.6.184. No abstract available. PMID 17213178
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Gupta N, Pinto LM, Morogan A, Bourbeau J. The COPD assessment test: a systematic review. Eur Respir J. 2014 Oct;44(4):873-84. doi: 10.1183/09031936.00025214. Epub 2014 Jul 3. PMID 24993906
- [Background] Karloh M, Fleig Mayer A, Maurici R, Pizzichini MMM, Jones PW, Pizzichini E. The COPD Assessment Test: What Do We Know So Far?: A Systematic Review and Meta-Analysis About Clinical Outcomes Prediction and Classification of Patients Into GOLD Stages. Chest. 2016 Feb;149(2):413-425. doi: 10.1378/chest.15-1752. Epub 2016 Jan 12. PMID 26513112
- [Background] Kon SS, Canavan JL, Jones SE, Nolan CM, Clark AL, Dickson MJ, Haselden BM, Polkey MI, Man WD. Minimum clinically important difference for the COPD Assessment Test: a prospective analysis. Lancet Respir Med. 2014 Mar;2(3):195-203. doi: 10.1016/S2213-2600(14)70001-3. Epub 2014 Feb 4. PMID 24621681
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Baker SEE, R. . How many qualitative interviews is enough? Expert voices and early career reflections on sampling and cases in qualitative research. National Centre for Research Methods. 2012.
- [Background] Ziebland S, McPherson A. Making sense of qualitative data analysis: an introduction with illustrations from DIPEx (personal experiences of health and illness). Med Educ. 2006 May;40(5):405-14. doi: 10.1111/j.1365-2929.2006.02467.x. PMID 16635119
- [Background] Joffe HaY, L., . Content and thematic analysis. Research methods for clinical and health psychology. California:. Sage. 2004:56-68.
- [Background] Ritchie J LJ, McNaughton Nicholls C, Ormston R. . Qualitative research practice: a guide for social science students and researchers. Sage. 2013.
- [Background] Johnson R, Waterfield J. Making words count: the value of qualitative research. Physiother Res Int. 2004;9(3):121-31. doi: 10.1002/pri.312. PMID 15560669